CLINICAL TRIAL: NCT06697782
Title: Clinical Study of Aprepitant and Ondansetron Monotherapy or Combination in the Treatment of Postoperative Nausea and Vomiting in Thyroid Carcinoma
Brief Title: Aprepitant and Ondansetron Monotherapy or Combination for Postoperative Nausea and Vomiting in Thyroid Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Shumin Dong, Clinical Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HN-PONV-ADR-01
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Ondansetron; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ondansetron group (Other): Patients in the ondansetron group received 8 mg of ondansetron orally 1 hour before anesthesia and twice at 8-hour intervals thereafter
  Interventions: Drug: Ondansetron 8mg
- Arepitant group (Other): Patients in the aprepitant group received 125 mg of aprepitant orally 1 hour before anesthesia and 80 mg orally once daily in the morning of postoperative days 2 and 3 (the day of the surgery was day 1)
  Interventions: Drug: Aprepitant 125 mg
- Combined treatment group (Experimental): Patients in the combined group received 125 mg of oral aprepitant plus 8 mg of ondansetron 1 hour before anesthesia, with ondansetron followed by two oral doses of the drug at 8-hour intervals, and 80 mg of aprepitant once daily in the morning on postoperative days 2 and 3 (the day of the surgery was day 1)
  Interventions: Drug: Ondansetron 8mg; Drug: Aprepitant 125 mg

INTERVENTIONS:
Drug: Ondansetron 8mg — Patients in the ondansetron group received 8 mg of ondansetron orally 1 hour before anesthesia and twice at 8-hour intervals thereafter
  Other Names: AD
  Arms: Combined treatment group; Ondansetron group
Drug: Aprepitant 125 mg — Patients in the aprepitant group received 125 mg of aprepitant orally 1 hour before anesthesia and 80 mg orally once daily in the morning of postoperative days 2 and 3 (the day of the surgery was day 1)
  Other Names: AR
  Arms: Arepitant group; Combined treatment group

SUMMARY:
The vast majority of patients treated prophylactically with "first-line" antiemetics in the 5-hydroxytryptamine (5-HT3) receptor antagonist class still have significant PONV. Combination therapies with different pharmacologic bases have the potential to reduce the incidence of PONV. This study is a multicenter, three-arm, prospective study to evaluate the efficacy and safety of aprepitant and ondansetron, monotherapy or in combination, in the prevention of nausea and vomiting after surgery for thyroid cancer.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is the most common complication after surgery, especially thyroidectomy, and the incidence of PONV can be as high as 80% without the administration of prophylactic antiemetics. Currently, available prophylactic interventions for PONV, especially monotherapy, lack universal efficacy. Combination therapy with a different pharmacologic basis has the potential to reduce the incidence of PONV. Previous studies using various 5-HT3 receptor antagonists in combination with aprepitant have shown promising results in reducing the incidence of PONV. The present study is a multicenter, three-arm, prospective study designed to evaluate the efficacy and safety of aprepitant and ondansetron, alone or in combination, in the prevention of postoperative nausea and vomiting in thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years;
2. Voluntary enrollment in the study and signing the informed consent form;
3. Diagnosed with thyroid cancer and needing surgical treatment;

Exclusion Criteria:

1. Patient has depression, history of chronic pain, insulin-dependent diabetes mellitus I or II, history of severe vomiting;
2. history of prior thyroid or neck surgery;
3. Cases in which surgery requiring sternotomy is anticipated;
4. History of long-term hormone use, period of immunosuppressive therapy;
5. pre-operative voice changes or laryngoscopic confirmation of vocal cord paralysis;
6. Pregnant or breastfeeding patients;
7. Patients who are allergic to any of the study medications;
8. Patients who have received any sedative, hypnotic, anxiolytic, opioid, steroid or other antiemetic medication within 24 hours prior to the procedure;
9. Patients taking or planning to take a combination of drugs such as rifampicin, carbamazepine, phenytoin or other drugs that strongly induce CYP3A4 activity;
10. patients with other malignant tumors;
11. Patients with hypothyroidism;
12. Participating or planning to participate in other clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Complete remission rate (CR rate) | Within 24 hours after surgery
  Complete remission rate (CR rate) without vomiting within 24h postoperatively and without resolution

SECONDARY OUTCOMES:
Complete remission rate (CR rate) | Within 48 hours after surgery
  Complete remission rate (CR rate) without vomiting within 48h postoperatively and without resolution
Rate of no vomiting | Within 24 and 48 hours after surgery
  Rate of no vomiting within 24h, 48h
Incidence of adverse events and serious adverse events | up to 24 weeks
  Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Detao Yin, M.D., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No